CLINICAL TRIAL: NCT04552938
Title: The Impact of Lymphaticovenous Anastomosis on Serum Profiling in Patients With Lymphedema
Brief Title: LVA on Serum Profiling in Patients With Lymphedema
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201800306B0
Record Dates: First submitted 2020-09-14; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2018-04

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients underwent supermicrosurgical LVA: Patients underwent supermicrosurgical LVA between June 2018 and May 2019.
  Interventions: Other: pre-LVA; Other: post-LVA

INTERVENTIONS:
Other: pre-LVA — Venous serum samples were collected from patients before LVA.
Other: post-LVA — Venous serum samples were collected from patients one-month after LVA.

SUMMARY:
The correlation between oxidative stress and increased lymphedematous limb volume lacks supporting evidence. Lymphedema patients are prone to cellulitis. This study aims to investigate the link between oxidative stress, limb volume, and cellulitis after supermicrosurgical lymphaticovenous anastomosis (LVA).

DETAILED DESCRIPTION:
In this study, we focused on the changes in serum antioxidant biomarkers before and after LVA, detected by isobaric tags for relative and absolute quantitation (iTRAQ)-based quantitative proteomic analysis, enzyme-linked immunosorbent assay (ELISA), and Oxidative Stress Panel Kit. For clinical correlation, magnetic resonance (MR) volumetry was implemented for precise lymphedematous limb volume measurements. Correlations were made between changes in oxidative stress, limb volume, and cellulitis before and after LVA.

ELIGIBILITY:
Inclusion Criteria:

* patients with lower limb lymphedema confirmed with lymphoscintigraphy
* unilateral lower limb lymphedema
* lymphedema duration > 2 years
* no active infection
* no prophylactic antibiotic use for at least one month before LVA
* no tumor recurrence or metastasis
* no consumption of antioxidants, such as vitamin E or ascorbic acid

Exclusion Criteria:

* Patients with upper limb and bilateral lower limb lymphedema

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Written informed consent was obtained from all patients. Between June 2018 and May 2019, 26 patients with lower limb lymphedema confirmed with lymphoscintigraphy were recruited. Patients with upper limb and bilateral lower limb lymphedema were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
the correlation between post-LVA volume reduction | 6 months after surgery
  The primary outcome was determined whether post-LVA volume reduction < 40%

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan